CLINICAL TRIAL: NCT00011440
Title: Markers of Pollutant Altered Allergic Responses
Brief Title: Pollutant Altered Allergic Responses
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 8077-CP-001
Record Dates: First submitted 2001-02-20; First posted 2001-02-21 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Allergic Rhinitis; Allergy
Keywords: Allergy; Air pollution; Lung function; Inflammation
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity; Inflammation

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
This study is designed to investigate whether exposure to particulate air pollution increases the allergic response to allergens. Research studies suggest that symptoms in individuals with allergies may be aggravated by exposure to particulate air pollution. We sought to experimental determine this by exposing human volunteers to combustion particles, a component of air pollution, and then challenge them with an allergen such as ragweed or oak tree pollen. Using biological tests we can measure whether the allergen response is magnified by prior particulate exposure.

DETAILED DESCRIPTION:
To study whether particulates enhance the allergic response, we chose the upper airway as a model of allergic inflammation and nasal lavage as a non-invasive method for obtaining samples. The nasal cavity is both an excellent model of allergic inflammation and provides an easily accessible site for study. We measured inflammatory cells and cytokines in the nasal lavage fluid. Our specific hypothesis was that particulate exposure prior to allergen challenge would enhance inflammatory cell recruitment and expression of inflammatory cytokines.

ELIGIBILITY:
Adult without a history of asthma or respiratory disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 1998-12; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard School of Public Health, Boston, Massachusetts, United States